CLINICAL TRIAL: NCT02256644
Title: CSP #575B - Genomics of Posttraumatic Stress Disorder Among Veterans
Brief Title: Genomics of Posttraumatic Stress Disorder in Veterans
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 575B
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Affymetrix Axiom Biobank chip, with technical specifications including "295K tag SNPs", "260K exomic content", "65K loss-of-function SNPs & INDELs", "25K psych content", and "23K eQTL markers".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Million Veteran Program (MVP) participants: Veterans who are currently enrolled in the Million Veteran Program.

SUMMARY:
Posttraumatic Stress Disorder (PTSD), as a common and serious mental health condition, affects about 25% of all military personnel that have served in combat. People suffering from PTSD may experience traumatic flashbacks, trouble sleeping, and problems in their relationships. This study is intended to help identify genes that influence and increase the risk of PTSD, to improve ways of detecting and treating the condition in the future.

Previous research has studied genes that increase the risk of PTSD, but none of these have included a Veteran-only population. The current study focuses on US Veterans, utilizing the VA Million Veteran Program (MVP) database of approximately 300,000 participants as of August 2014. In this context, participants with PTSD are referred to as "cases" and Veterans without PTSD are referred to as "controls."

This project will be done in three stages. The first stage will look at MVP-obtained data and electronic health record (EHR) data to implement methods for identifying combat-exposed case patients with PTSD and combat-exposed control patients without PTSD. The second stage will assemble and validate a study population of 20,000 participants "including 10,000 combat-exposed Veterans with PTSD as cases and 10,000 combat-exposed Veterans without PTSD as controls. The third stage will conduct genetic analyses ("genotyping") comparing the cases to controls, to identify genes associated with increased risk of developing the condition.

DETAILED DESCRIPTION:
Background and Objectives

Posttraumatic stress disorder (PTSD) is a severe, sometimes disabling, anxiety disorder that can develop after a potentially traumatic event involving actual or threatened death, serious injury, or sexual violation. The diagnosis of PTSD requires symptoms for at least one month from three categories: re-experiencing, avoidance, and increased arousal. In contrast to an acute response to trauma, the stress reactions of persons who develop PTSD do not resolve quickly; symptoms can last for long periods of time and may increase in severity.

The rate of PTSD (and consequent disability) is especially high among combat-exposed military Veterans. Studies of Vietnam combat veterans have consistently found a lifetime PTSD prevalence of 25-30% of men, although rates of persistent/chronic PTSD have been somewhat lower (15-20%). Studies of OEF/OIF Army personnel have reported rates of PTSD in the 10% to 15% range following deployment (Thomas et al 2010). These rates are much higher than the rate of PTSD in the general US population, estimated to be about 6.8% (Kessler et al 2005).

PTSD has been shown to be influenced genetically, and previous work has identified several possible genes that increase the risk of PTSD. Although several genomewide association studies (GWASs) have been conducted, the corresponding statistical power has been modest, and none included a Veteran-only population. The proposed study will address those deficiencies by conducting a well-powered case-control GWAS study in a large sample of US Veterans with PTSD as "cases" and psychiatrically-healthy Veterans as "controls."

Preliminary Data and Research Design

The study will use a case-control design nested within the VA Million Veteran Program (MVP), with genotype as the exposure variable and PTSD diagnosis (yes/no) as the outcome variable. The pool of potential PTSD cases will be identified initially based on self-report of a PTSD diagnosis on a previously completed self-report questionnaire collected in MVP, or evidence of a PTSD diagnosis in the VA electronic health record (EHR). Specific validation procedures will narrow the pool to confirmed PTSD cases and controls. Based on available MVP and VA EHR data, the investigators estimate a currently available source population of more than 11,000 confirmed PTSD cases among the approximately 145,000 MVP enrollees to date. By the time this project gets underway, the number of available cases (and controls) will be even higher, due to ongoing enrollment into MVP.

Laboratory Methods and Statistical Analyses

This PTSD GWAS will compare 10,000 combat-exposed Veterans with PTSD to 10,000 combat-exposed controls. A to-be-selected microarray (see narrative) will be employed that contains approximately 245K genomewide association markers, 250K exonic markers and INDELs, 70K novel loss-of-function SNPs and INDELs, and 115K "custom" markers. Genotypes will be imputed to approximately 1KG for statistical analysis, and up to 50 putatively-associated SNPs that are initially imputed will be genotyped directly in the same sample.

Anticipated Results and Relevance

Genetic loci affecting combat-related PTSD risk and resilience will be identified, providing important information to inform therapeutic targets related to prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Combat-exposed Veterans who participated in the Million Veteran Program.

Exclusion Criteria:

* schizophrenia
* bipolar disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators expect 70-80% European-American (EA) and 20-30% African American (AA) in the current study
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
PTSD diagnosis | 2 years
  The study will use a case-control design nested within the VA Million Veteran Program (MVP), with genotype as the exposure variable and PTSD diagnosis (yes/no) as the outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD MPH, Study Chair — VA San Diego Healthcare System, San Diego, CA; Joel Gelernter, MD, Study Chair — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Austin-Zimmerman I, Levey DF, Giannakopoulou O, Deak JD, Galimberti M, Adhikari K, Zhou H, Denaxas S, Irizar H, Kuchenbaecker K, McQuillin A; Million Veteran Program; Concato J, Buysse DJ, Gaziano JM, Gottlieb DJ, Polimanti R, Stein MB, Bramon E, Gelernter J. Genome-wide association studies and cross-population meta-analyses investigating short and long sleep duration. Nat Commun. 2023 Sep 28;14(1):6059. doi: 10.1038/s41467-023-41249-y. PMID 37770476
- [Derived] Radhakrishnan K, Aslan M, Harrington KM, Pietrzak RH, Huang G, Muralidhar S, Cho K, Quaden R, Gagnon D, Pyarajan S, Sun N, Zhao H, Gaziano M, Concato J, Stein MB, Gelernter J. Genomics of posttraumatic stress disorder in veterans: Methods and rationale for Veterans Affairs Cooperative Study #575B. Int J Methods Psychiatr Res. 2019 Mar;28(1):e1767. doi: 10.1002/mpr.1767. Epub 2019 Feb 14. PMID 30767326
- See also: Related Info — http://www.research.va.gov/programs/csp/csp575B.cfm